CLINICAL TRIAL: NCT00628758
Title: A Comparison of Symbicort® Single Inhaler Therapy (Symbicort Turbuhaler® 160/4.5mg, 1 Inhalation Two Times a Day (b.i.d.) Plus as Needed) and Conventional Best Practice for the Treatment of Persistent Asthma in Adults a -26-week, Randomized, Open-label, Parallel-group, Multicentre Study
Brief Title: A Comparison of Symbicort® Single Inhaler Therapy and Conventional Best Practice for the Treatment of Persistent Asthma
Acronym: PASSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00016
Record Dates: First submitted 2008-01-10; First posted 2008-03-05 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Symbicort; Turbuhaler; Persistent Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort (Experimental): Symbicort Single Inhaler Therapy ( Turbuhaler 160/4.5 microgram, 1 inhalation bid + as needed)
  Interventions: Drug: Symbicort TBH - Turbuhaler
- Conventional BP (Experimental): Conventional Best Practice for Treatment of Asthma
  Interventions: Drug: beta-II-agonist, inhale steroid

INTERVENTIONS:
Drug: Symbicort TBH - Turbuhaler — Symbicort Single Inhaler Therapy ( Turbuhaler 160/4.5 microgram, 1 inhalation bid + as needed)
  Arms: Symbicort
Drug: beta-II-agonist, inhale steroid — Salbulin inh. 200-400 dosage 100 microgram (mcg)/dosage Salbutamol Sustained Release(SR)capsule 4 mg/8 mg Salbutol tablet (tb) 2 mg Salbutol forte syrup 2 mg/5 ml Ventolin tb, syrup, intravenous(IV),5mgx10 ampule(amp) Ventolin inhaler (inh) 200 dosage, 100 mcg/dosage Ventolin nebul 2.5 mg Volmax tb 4 mg/8 mg Vent-o-sal inh 100 mcg/200 dosage Combivent inh 100 mcg/dosage Combivent neb 2.5 mg/dosage Bricanyl tb 2.5 mg Bricanyl durules ret tb 5 mg Bricanyl syrup 30mg Bricanyl inhaler 0.25 mg/dosage, 400 dosage Bricanyl turbuhaler 0.5 mg/dosage, 200dosage
  Other Names: Astmerol inh 25 mcg/dosage, 60-120 dosage; Astmerol maksihaler 50 mcg/dosage, 28-60 dosage; Serevent diskus 50 mcg/dosage, 60 dosage; Serevent inh 25 mcg/dosage, 60 dosage; Foradil inh kap 12 mcg/dosage, 60 caps; Foradil inh 12 mcg/dosage, 50-100 dosage; Foradil combi 200 mcg; Foradil combi 400 mcg; Oxis turbuhaler 4.5-9 mcg/dosage, 60 dosage; Ventofor 12mg/60 inh.caps; Seretide disc 100-250-500 mcg/dosage 60 dosage; Symbicort 160/4.5 mcg/60-120 dosage, 320/9mcg/60 dosage
  Arms: Conventional BP

SUMMARY:
The primary objective is to compare the efficacy of Symbicort Single inhaler Therapy with treatment according to conventional best practice in adult patients with persistent asthma.

DETAILED DESCRIPTION:
A secondary objective is to collect safety data for treatment wtih Symbicort Single inhaler Therapy in adult patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form. If the patient cannot read and write, verbal consent from the patient is required.
* Ability to read and write in Turkish
* Female or male outpatients aged 18 years
* Minimum of 3 months history of asthma, diagnosed according to the American Thoracic Society (ATS) definition
* Prescribed inhaled glucocorticosteroid (GCS) at a dose of 320mg/day and within the approved label for the relevant drug during the last 3 months prior to Visit 1
* Either: daily maintenance treatment with both inhaled GCS and long-acting b2-agonist (LABA) or daily treatment with inhaled GCS alone (i.e. without LABA); and a history of suboptimal asthma control the month prior to enrollment as judged by the investigator; and use of 3 Peak Expiratory Flow inhalations ofas needed medication for symptom relief during the last 7 days before enrollment

Exclusion Criteria:

* Previous treatment with Symbicort Single inhaler Therapy
* Use of any b-blocking agent, including eye drops
* Use of oral GCS as maintenance treatment
* Known or suspected hypersensitivity to study therapy or excipients
* A history of smoking 10 pack years
* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator
* Any significant disease or disorder, which, in the opinion of the investigator, may put the patient at risk because of participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Misirligil, Principal Investigator — Ankara Univ. Med. Fac, Chest Disease Dept
Locations (15):
- Turkey (Türkiye) (15):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Denizli
  - Research Site, Diyarbakır
  - Research Site, Edirne
  - Research Site, Eski?ehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Malatya
  - Research Site, Manisa
  - Research Site, Mersin
  - Research Site, Samsun
  - Research Site, Zonguldak

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FSI: LSI: LSO: Center type: Research and Training Host, Chest Medicine and Internal Medicine 23 Clinics. Number of enrolled subjects: 432, randomized: 430, completed patients: 344 ( Arm A:165, Arm B 179)
Groups:
- Symbicort: Symbicort Single Inhaler Therapy ( Turbohaler 160/4.5 microg, 1 inh bid + as need)
Period: Overall Study
Arm/Group | Symbicort | Conventional BP
Started | 209 | 221
Completed | 165 | 179
Not Completed | 44 | 42
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 5 | 1
Not completed — Lost to Follow-up | 25 | 31
Not completed — Pregnancy | 2 | 2
Not completed — Investigator Moved | 3 | 0
Not completed — Treatment Failure | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort | Conventional BP | Total
Number analyzed (Participants) | 209 | 221 | 430
Age Continuous [Mean (Standard Deviation); unit: years] | 44.28 (12.09) | 45.17 (12.71) | 44.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 179 | 336
  Male | 52 | 42 | 94

OUTCOME MEASURES:

1. Primary Outcome: Time to First Severe Asthma Exacerbation
Description: Time to severe exacerbation among patients
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Symbicort: Symbicort Single Inhaler Therapy ( Turbohaler 160/4.5 microgram (microg), 1 inh bid + as need)
- Conventional Best Practice (BP): Conventional Best Practice for Treatment of asthma
Arm/Group | Symbicort | Conventional Best Practice (BP)
Number analyzed (Participants) | 209 | 221
days | 120.3 (47.0) | 103.7 (32.7)

2. Secondary Outcome: Number of Severe Asthma Exacerbations
Description: Total number of severe asthma exacerbations per treatment group
Time Frame: 26 weeks
Measure: Number; unit: Severe Exacerbations
Arm/Group | Symbicort | Conventional BP
Number analyzed (Participants) | 209 | 221
Severe Exacerbations | 10 | 10

3. Secondary Outcome: Change in Standardised Asthma Quality of Life Questionnaire (AQLQ(S)) Score
Description: Quality-of-Life assessment; grouped in four domains;activity limitation, symptoms, emotional function and exposure to environmental stimuli, using with a scale from 1 to 7 where 1 represents the greatest possible impairment and 7 represents the least impairment.
Time Frame: Baseline and 26 weeks
Population: ITT analysis was performed. Being in line with the analysis description population and due to the description of the variable. This patient-reported outcome variable could only be calculated for patients who have baseline and visit 4 AQLQ data. The AQLQ was not filled in by all enrolled patients.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort | Conventional BP
Number analyzed (Participants) | 146 | 154
Units on a scale | 3.98 (1.12) | 3.97 (1.15)

4. Secondary Outcome: Mean Use of As-needed Medication Per Day During Treatment Period
Description: Mean use of as-needed medication per day during treatment period
Time Frame: Daily recording during the treatment period of 26 weeks
Population: ITT analysis was performed. Being in line with the analysis description population and due to description of the variable which was based on the patient's estimate, this variable could only be calculated of the patients who had recorded at least one estimate on their dairies they had been asked to return to the investigator at the study visits.
Measure: Mean (Standard Deviation); unit: inhalations per day
Arm/Group | Symbicort | Conventional BP
Number analyzed (Participants) | 178 | 193
inhalations per day | 0.91 (7.6) | 0.68 (5.7)

ADVERSE EVENTS:
Arm/Group | Symbicort | Conventional BP
Serious Adverse Events (participants affected / at risk) | 2/209 | 2/221
Other Adverse Events (participants affected / at risk) | 0/209 | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=209) | Conventional BP (N=221)
Cardiac Arrest (Cardiac disorders) | 1 | 0
Lower Limb Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No